CLINICAL TRIAL: NCT03334578
Title: The Use of Gastrografin to Help Alleviate Bowel Obstruction Related to Poor Bowel Motility in Gastroschisis Patients.
Brief Title: The Use of Gastrografin to Help Alleviate Bowel Obstruction in Gastroschisis Patients.
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of recruitment
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 109470
Record Dates: First submitted 2017-10-30; First posted 2017-11-07 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Gastroschisis; Bowel Obstruction; Birth Defect
MeSH Terms: conditions — Gastroschisis; Intestinal Obstruction; Congenital Abnormalities | interventions — Diatrizoate Meglumine; Diatrizoate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Drug: Gastrografin (Experimental): Patient will receive 30ml of Gastrografin (diluted at 1:3 ratio with water) as recommended by the manufacturer for a single dose in our population. The dose will be given via the nasogastric tube, which will then be clamped for 1 hour. Gastrografin will only be given if there is evidence of a bowel obstruction. Additionally, Gastrografin will only be given when the patient is hemodynamically stable, not receiving any inotropes, and off of invasive respiratory support. Once administered the patient will receive an x-ray at 48 hours. If Gastrografin can be viewed past the obstruction than another dose of Gastrografin (30ml at 1:3 dilution ratio with water via NG tube) can be given. If gastrografin is not viewed past the obstruction than another dose will not be given.
  Generic name: Diatrizoate Meglumine, Diatrizoate Sodium
  Interventions: Drug: Gastrografin
- Control: Standard care (No Intervention): This group will be recruited from an ongoing observational study at our centre. The patients in this group have all received the standard care for treating gastroschisis and any potentially associated bowel obstruction. They have not received Gastrografin. They will be recruited between May 2010 and May 2019.

INTERVENTIONS:
Drug: Gastrografin — Gastrografin group
  Other Names: Diatrizoate Meglumine; Diatrizoate Sodium
  Arms: Drug: Gastrografin

SUMMARY:
This study will investigate the use of a drug called Gastrografin to aid in bowel mobility for paediatric patients who have undergone gastroschisis surgery. Gastroschisis is an abdominal wall birth defect where the bowel protrudes through a small opening beside the umbilicus. In these patients, the bowel is often less mobile due to its exposure outside of the body during fetal development. It is common for the bowel to be swollen and matted, which decreases motility and makes it increasingly difficult for the baby to have normal bowel function. Administering Gastrografin facilitates the entry of water into the intestines and bowel, which is thought to aid in bowel function and motility. This study will compare gastroschisis patients who received Gastrografin to gastroschisis patients collected as part of an ongoing observational study at our centre who did not receive Gastrografin.

DETAILED DESCRIPTION:
Gastroschisis is a congenital birth defect where the fetal abdominal organs (typically the intestines) protrude through a defect in the abdominal wall, just to the right of the umbilicus. For babies born with gastroschisis, once the child is considered to be hemodynamically stable, surgery can be performed to reduce the bowel back into the abdominal cavity. Typically the use of immediate or delayed closure of the abdominal cavity is based on the child's condition, the size of the defect and the amount of bowel that is outside of the abdominal cavity. Most often the placement of a surgical silo can enable gentle reduction of the contents back into the abdomen, allowing for surgical closure of the abdominal opening. Due to the exposure of the baby's bowel to the mother's amniotic fluid during fetal development in the womb, the bowel can become matted and edematous. This often prevents normal bowel motility and can act as a functional bowel obstruction, making it difficult for the baby to pass the meconium at birth or initiate normal stooling. In more severe cases fibrous bands of tissue can develop along the bowel, causing a mechanical bowel obstruction that requires operative management.

Most often these functional and mechanical obstructions are treated conservatively/non-surgically for upwards of 6 weeks (i.e., nasogastric (NG) tube decompression, nothing per mouth (NPO) and intravenous (IV) fluids). If resolution has not occurred after this time period the parents/guardians can request elective surgery, after 6 weeks and when the baby is stable, to help resolve the obstruction. The waiting period between surgical closure of the contents back into the abdomen and the initiation of feeding is a critical time as the baby typically experiences bilious vomiting and an aversion to feeding which can impact their physical development.

Gastrografin is a hyperosmolar water-soluble contrast agent that has a therapeutic benefit of stimulating the mobility of the intestines and drawing water from the bowel walls into the lumen. Gastrografin is used as a therapeutic agent in a number of obstructive clinical scenarios including small bowel obstruction in paediatric and adult populations and in meconium ileus and meconium plug syndrome in the neonate. Patients with gastroschisis have a similar symptomology as the previously mentioned patients and therefore may benefit from the therapeutic use of Gastrografin. This study will be the first known study to examine the use of Gastrografin in this population.

This is a single centre open-labeled clinical trial that is investigating a new indication for an approved prescription drug by the FDA and Health Canada. The drug used in this study is called Gastrografin, it is marketed as a radiopaque contrast agent that has a mild laxative effect due to its osmolarity. This study looks to further study this laxative property to alleviate bowel obstructions in babies born with gastroschisis. This study has two parts: first, the Gastrografin group will be recruited between October 1st, 2017 and September 30th, 2019 as part of this clinical trial. Second, the Gastrografin group will be linked to a cohort of gastroschisis patients who have been collected as part of an ongoing approved observational study at Western University (REB# 2436) between May 1st, 2010 and May 1st, 2019. The ongoing study is part of the Canadian Neonatal Network (CNN) and the Canadian Pediatric Surgery Network (CAPSNET). The May cut-off date is required because that is when the data collected at our site is uploaded and made available for research purposes. The patients in the Gastrografin group will be matched to the non-Gastrografin group on age, birth weight, sex, and the Score for Neonatal Acute Physiology (SNAP) at 12 hours after admission, to ensure that the groups are representative of one another. Since these babies are born with gastroschisis and are treated immediate from birth, there is no pre-screening visit and once consent is obtained from the caregivers the baby will be entered into the Gastrografin protocol. The study period will last from admission to discharge, there are no follow-up time points in this study where data will be collected. Patients will be seen in clinic for follow-up as per standard procedure for gastroschisis.

ELIGIBILITY:
Inclusion Criteria:

- Diagnosis of gastroschisis

Exclusion Criteria:

* Gestational age less than 32 weeks
* Birth weight less than 1500 grams
* Definitive bowel atresia based on physician diagnosis

Ages: 32 Weeks to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2018-08-03 (Actual); Primary Completion 2020-12-17 (Actual); Study Completion 2020-12-17 (Actual)

PRIMARY OUTCOMES:
Time to Start Feeds | From the date of admission at the hospital to the date feeding is initiated, assessed up to 6 months
  The length of time in days from admission/birth to initiate feeding.
Time to Reach Full Feeds | From the date feeding was initiated to the date when the patient reaches full feeds (defined clinically- varies based on individual patient), assessed up to 6 months
  The length of time in days from when feeding was initiated to when baby is considered fully fed

SECONDARY OUTCOMES:
Length of Hospital Stay | upwards of 6 months based on receiving standard care
  The time between admission/birth to discharge
Complication Rate | Up of 6 months
  The rate of other such complications associated with gastroschisis or Gastrografin during hospital stay
Operative rate | Up to 6 months
  The rate of elective surgeries in both groups to treat bowel obstruction during hospital stay

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital, London Health Sciences Centre, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No